CLINICAL TRIAL: NCT00547365
Title: Therapeutic Potential of Human Immune Globulin Intravenous (IGIV) in Patients With Cardiac-Associated Light Chain (AL) Amyloidosis
Brief Title: Human Immune Globulin in Treating Patients With Primary Amyloidosis That is Causing Heart Dysfunction
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Tennessee (Other)
Responsible Party: Principal Investigator, Alan Solomon, Professor of Medicine, University of Tennessee
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000572104; BRCC-BHS-06127 (Other: Baxter); UTCI-2645 (Other: Baxter)
Record Dates: First submitted 2007-10-19; First posted 2007-10-22 (Estimated); Results first posted 2013-09-19 (Estimated); Last update posted 2013-09-19 (Estimated); Status verified 2013-09

CONDITIONS: Multiple Myeloma; Plasma Cell Neoplasm
Keywords: primary systemic amyloidosis
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell; Immunoglobulin Light-chain Amyloidosis | interventions — Immunoglobulins, Intravenous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Human immune globulin intravenous (IGIV) (Experimental): Analyze the therapeutic potential of human immune globulin intravenous (IGIV) when given to patients with cardiac-associated AL amyloidosis
  Interventions: Biological: Human immune globulin intravenous (IGIV)

INTERVENTIONS:
Biological: Human immune globulin intravenous (IGIV) — Analyze the therapeutic potential of human immune globulin intravenous (IGIV) when given to patients with cardiac-associated AL amyloidosis

SUMMARY:
RATIONALE: Antibodies, such as human immune globulin, can block the growth of abnormal cells in different ways. Some block the ability of abnormal cells to grow and spread. Others find abnormal cells and help kill them or carry cell-killing substances to them. Giving human immune globulin may be effective in treating patients with primary amyloidosis that is causing heart dysfunction.

PURPOSE: This phase I/II trial is studying the side effects and best dose of human immune globulin and to see how well it works in treating patients with primary amyloidosis that is causing heart dysfunction.

DETAILED DESCRIPTION:
OBJECTIVES:

* Establish the maximum tolerated dose of human immune globulin intravenous (IGIV) given weekly for the first 3 months and then bi-weekly for 9 additional months in patients with cardiac-associated primary light chain-associated (AL) amyloidosis.
* Determine the safety, pharmokinetics, and therapeutic efficacy as evidenced by titers of serum fibril-reactive immunoglobulin G (IgG) antibodies pre- and post-IGIV infusions.
* Demonstrate stable or improved organ function.

OUTLINE: Patients receive human immune globulin IV (IGIV) once weekly for 3 months and then once biweekly for 9 months, for a total of 12 months in the absence of disease progression or unacceptable toxicity.

Patients undergo blood sample collection to measure serum anti-fibril antibody titers pre- and post- IGIV infusion for assessing safety and response to treatment.

ELIGIBILITY:
Inclusion criteria:

* Confirmed diagnosis of cardiac-associated primary (AL) amyloidosis based on accepted clinical and laboratory criteria
* Patients must have heart involvement as evidenced by elevated serum brain natriuretic peptide (BNP), troponin levels, and/or 2D echocardiography evidence of a thickened intraventricular septum (IVS).
* Life expectancy > 3 months
* Prior or concurrent chemotherapy or other drug-based anti-AL regimes allowed

Exclusion criteria:

* Non-AL amyloidosis
* New York Heart Association (NYH) class IV heart disease
* Significant comorbidity (e.g., uncontrolled infection, diabetes, or other serious illnesses)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-10; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan Solomon, MD, Study Chair — St. Mary's Medical Center
Locations (2):
- United States (2):
  - Baptist Regional Cancer Center at Baptist Riverside, Knoxville, Tennessee
  - St. Mary's Medical Center, Powell, Tennessee

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Overall study length - 2007-2011; Location - medical clinic
Pre-assignment Details: Patients with primary light-chain (AL)-associated amyloidosis that caused heart dysfunction were on study.
Groups:
- Human Immune Globulin Intravenous (IGIV): The therapeutic potential of human immune globulin intravenous (IGIV)was evaluated in patients with cardiac-associated AL amyloidosis. Patients received, via intravenous infusion, 30-40 gm of IGIV (depending on body weight) weekly for 3 months and then every other week for the next 9 months.The total time to complete the study was ~1 yr.
Period: Overall Study
Arm/Group | Human Immune Globulin Intravenous (IGIV)
Started | 10
Completed | 2
Not Completed | 8
Not completed — Physician Decision | 1
Not completed — Lost to Follow-up | 1
Not completed — Protocol Violation | 2
Not completed — death (not related to study) | 4

BASELINE CHARACTERISTICS:
Population: Patients with cardiac-dominant AL amyloidosis, as determined from standard clinical tests (IVS, BNP),were entered on study.
Arm/Group | Human Immune Globulin Intravenous (IGIV)
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Tolerance for Human Immune Globulin Intravenous (IGIV), as Reflected by the Number and Severity of Toxicity Incidents Occurring in Ten Patients Receiving at Least One Infusion of IGIV.
Time Frame: Up to 1 year
Population: All patients who had at least one infusion of human immune globulin intravenous.
Measure: Number; unit: events
Groups:
- Human Immune Globulin Intravenous (IGIV): Immune globulin intravenous (IGIV) was administered to patients with cardiac-dominant AL amyloidosis in order to determine its therapeutic potential or possible toxicity when given to subjects weekly for 3 months and then every other week for the next 9 months. Response was evaluated by changes in serum anti-fibril antibody levels, changes in BNP (B-type natriuretic peptide) levels and IVS (interventricular septum) thickness.
Arm/Group | Human Immune Globulin Intravenous (IGIV)
Number analyzed (Participants) | 10
events | 0

2. Primary Outcome: Clinical Response of Patients With Cardiac-dominant AL Amyloidosis Given Human Immune Globulin Intravenous (IGIV)
Description: Positive clinical response was defined by improvement in heart function in participating patients with cardiac-dominant AL amyloidosis, as demonstrated by increased serum anti-fibril immunoglobulin G (IgG) antibody levels and reduction (or no evident progression) in amyloid burden.
Time Frame: Up to 1 year
Population: Two of ten patients with AL cardiac involvement who received IGIV infusions were analyzed (other eight individuals were removed from study before completion due to death/conditions unrelated to IGIV, loss to follow-up, or physician decision).
Measure: Number; unit: participants with positive response
Groups:
- Human Immune Globulin Intravenous (IGIV): Human immune globulin intravenous (IGIV) was infused into 10 patients with cardiac-associated AL amyloidosis and its therapeutic potential evaluated through measurement of serum anti-fibril IgG antibody levels, as well as amyloid burden, pre- and post-administration.
Arm/Group | Human Immune Globulin Intravenous (IGIV)
Number analyzed (Participants) | 2
participants with positive response | 1

ADVERSE EVENTS:
Groups:
- Human Immune Globulin Intravenous (IGIV): Therapeutic potential of human immune globulin intravenous (IGIV)in patients with cardiac-associated AL amyloidosis
Arm/Group | Human Immune Globulin Intravenous (IGIV)
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No